CLINICAL TRIAL: NCT02170285
Title: Enhancing Developmental Motor Plasticity After Perinatal Stroke With Transcranial Direct Current Stimulation
Brief Title: Enhancing Motor Plasticity After Perinatal Stroke Using tDCS
Acronym: tDCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Adam Kirton, Associate Professor, Pediatrics and Clinical Neurosciences, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: E24720
Record Dates: First submitted 2014-06-16; First posted 2014-06-23 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Perinatal Stroke; Cerebral Palsy
Keywords: perinatal stroke; hemiparetic cerebral palsy; brain stimulation; tDCS; constraint-induced movement therapy; hand arm bimanual intensive therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional tDCS (Experimental): The primary intervention will be cathodal (inhibitory) tDCS (see below).
  Interventions: Device: Interventional TDCS
- Sham tDCS (Sham Comparator): Sham subjects will undergo exactly the same tDCS protocol as outlined above. This includes the initial stimulation sequence, generating the initial transient scalp sensations identical to the treatment group. The stimulator will be programmed by the technologist to automatically ramp down to off over 30 seconds after 120 seconds of stimulation.
  Interventions: Device: Sham TDCS

INTERVENTIONS:
Device: Interventional TDCS — The primary intervention will be cathodal (inhibitory) tDCS over non-lesioned M1. This will be targeted using TMS baseline mapping data and neuronavigation (Brainsight2, Rogue Research, Montreal) individualized to the subjects MRI. Soft, replaceable 25cm2 electrodes will be placed over clean, dry scalp with the cathode over marked M1 and the reference electrode over contralateral forehead/orbit consistent with standard protocols. The current-controlled DC stimulator (neuroConn GmbH, Ilmenau, GE) will be turned up slowly over 30 seconds to the treatment current of 1.0 mA. TDCS will be administered each day during the first 20 minutes of the 90 minute therapy session. Child, family, and both treating and measuring occupational therapists are blinded to treatment allocation.
  Other Names: DC stimulator (neuroConn GmbH, GE)
  Arms: Interventional tDCS
Device: Sham TDCS — Sham subjects will undergo exactly the same tDCS protocol as outlined above. This includes the initial stimulation sequence, generating the initial transient scalp sensations identical to the treatment group. The stimulator will be programmed by the technologist to automatically ramp down to off over 30 seconds after 120 seconds of stimulation.
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to test tDCS (transcranial direct current stimulation), a type of non-invasive brain stimulation, to determine whether it can improve motor function in children with perinatal stroke and hemiparesis. Children 6-18 years with imaging-confirmed perinatal stroke and functional motor impairment will be recruited. Children will be randomized (1:1) to receive sham or tDCS (20 minutes daily) during daily intensive, goal-directed motor learning therapy (90 minutes). Motor outcomes will be repeated at baseline, 1 week, and 2 months.

Aim 1: Establish the ability of tDCS to safely enhance motor learning in children with perinatal stroke.

Hypothesis 1: tDCS is safe and well tolerated in children.

Hypothesis 2: Contralesional, cathodal tDCS increases motor functional gains measured by AHA at 2 months in children with perinatal stroke.

DETAILED DESCRIPTION:
Methods details not included elsewhere

Study: Randomized, sham-controlled, double blind, phase II clinical trial.

Patient Population. All children will be recruited through the Alberta Perinatal Stroke Project (APSP); a large population-based perinatal stroke research cohort based at Alberta Children's Hospital and directed by the PI. Prospective APSP ascertainment since 2007 is combined with retrospective enrolment (1992-2007) with comprehensive International Classification of Disease codes (ICD-9, ICD-10)237 and institutional databases. These are fully characterized patients with confirmed diagnosis by modern neuroimaging assessed in person in standardized APSP clinics. Recruitment will occur randomly from the population of all children meeting the criteria below.

Inclusion/exclusion criteria - see below

Data Collection and Management. Candidate APSP families will be contacted with review of consent/assent forms. Families residing outside Calgary will have equal opportunity to participate through existing APSP support systems. All complimentary data from existing studies is extractable from the APSP database (demographics, imaging, risk factors, outcomes).13 Neuroimaging data will be managed through the ACH Pediatric Neuroimaging Laboratory according to institutional protocols. Neurophysiology data will be collected at the ACH Pediatric TMS Laboratory and securely stored centrally.107 The institutional Clinical Research Unit is a database management unit designed for clinical research and currently houses all APSP studies and trials. The research database platform encompasses data capture utilities, management tools, and security measures (Health Canada-compliant). Methods will adhere to the CONSORT guidelines and the study will be registered prior to consent of the first patient (www.clinicaltrials.gov).

Intensive Motor Learning (all subjects). An evidence-based approach to upper extremity motor learning therapy in children with hemiparetic CP will be employed. Protocols have been designed by expert pediatric neurorehabilitation and occupational therapy co-investigators based on best available evidence. All children will participate in the same child-centered, age-appropriate, goal-directed, peer supported motor learning program. Designed as an "after school program" to optimize efficiency, children will attend our hospital for 10 consecutive weekdays over 2 weeks. Each session begins with a 30 minute social snack activity, providing the opportunity for peer social interactions and "recharging" from the school day while engaging their affected extremity in functional activity. Each subject then enters 90 minutes of goal-directed (see COPM in outcome measures) motor learning therapy with an individualized occupational therapist.

Week 1 will employ constraint induced movement therapy (CIMT) according to current practice guidelines. Each child will be custom fit with a removable, bivalved cast that will be worn throughout all therapy sessions. Week 2 will transition to intensive bimanual therapy to integrate gains into more practical bimanual functions. Intensive bimanual therapies are now evidence-based, safe, valid, and effective motor learning strategies in children with hemiparetic CP. Efficacy appears equal to CIMT but the absence of constraint facilitates functional bimanual motor learning and removes the complications of casting. Bimanual tasks will be graded and selected according to relative function with increasing complexity across the relevant spectrum (e.g. passive assist to active manipulator). Tasks will be both symmetrical and asymmetrical, geared to age-appropriate activities of daily living and individual interests, and include active patient participation. Following the acute 10 day intervention, all children receive a structured home program based on the same principles with ongoing therapist support, surveillance, and documentation for 2 months.

Randomization and blinding. Children will be randomized 1:1 to tDCS or sham. The study statistician will perform the randomization based on study number only, being blinded to all subject details. Allocation will then be communicated to the study PI and tDCS neurophysiologist only. The subject, parents, measuring and treating occupational therapists, and all other study members will be blinded to treatment allocation. The neurophysiologist will then program each subjects tDCS unit accordingly. All will experience identical ramp-up of current to 1mA over 30 seconds and maintained stimulation for 120 seconds. Those randomized to treatment will have the same current maintained for 20 minutes during therapy. The tDCS units of those randomized to sham will automatically ramp-down gradually to off over 60 seconds following the initial 120 seconds of stimulation. These sham procedures are well validated in adult tDCS trials. Blinding effectiveness will be evaluated.

Intervention: TDCS - see below.

Outcome measures - see below

Interim Safety Analysis. Any possible major side effects will be immediately reported to the IRB per policy. Minor side effects will be tracked by the safety outcomes specified. An interim safety analysis will be performed after the first 2 camps (12 subjects) to ensure no decrease in hand function has occurred in association with contralesional tDCS. This will be evaluated by comparing change in affected (AHA, MA) and unaffected (GS, PS, BB) hands at both 1 week and 2 months between tDCS and sham populations.

Sample Size. Variables were extrapolated from the most relevant literature, our previous studies in the same population, and personal communication with AHA creators. Smallest detectable difference for the AHA is estimated at 0.97 logit units or approximately 5 logit-based AHA units. Our previous trial in the same population found the proportion achieving this change was approximately 25% with CIMT alone compared to 65% receiving both CIMT and contralesional brain stimulation (rTMS). Therefore, for the primary hypothesis that tDCS improves AHA gains at 2 months, significance level alpha=0.05, power of 90%, and no drop-outs (100% completion in previous trials), 24 patients (12 per group) will be required. This is comparable or larger than most pediatric CP trials and positive tDCS and rTMS adult stroke trials.

Statistical Analysis. Co-investigator expertise in statistical methods (AN) and clinical trial methodology (MH) are established. Primary analysis will examine change in AHA and other outcome variables from baseline to final outcome at 2 months using simple ANOVA. Secondary analysis will explore effects of time and severity using repeated measures ANCOVA with deficit severity as a covariable to examine interactions across treatment groups (tDCS, sham). Safety outcomes will compare changes in unaffected hand function (as above), adverse event rates (tDCS vs sham) using Chi-square/Fisher exact and Mann-Whitney tests. Association between treatment group and subject's estimation of treatment received will be determined to evaluate sham effectiveness (Chi-square/Fisher exact). The sample is not large enough for multivariable modelling. Analysis will be intention-to treat.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic hemiparetic CP (Pediatric Stroke Outcome Measure (PSOM) >0.5) AND Manual Abilities Classification System (MACS) grade I-IV AND child/parent perceived limitations
2. Clinical and MRI-confirmed perinatal stroke syndrome (NAIS, APPIS, PVI)
3. Active wrist extension >20 degrees, finger extension >10 degrees
4. Can lift the affected arm 15 cm above a table surface and grasp light objects
5. Term birth (>36 weeks) and current age 6 - 18 years
6. Informed consent

Exclusion Criteria:

1. Other neurological disorder not related to perinatal stroke
2. Multifocal perinatal stroke
3. Severe hemiparesis (no voluntary contraction in paretic hand, MACS level V)
4. Severe spasticity in the affected limb (Modified Ashworth Scale >3)
5. Severe developmental delay or other inability to comply with study protocol
6. Unstable epilepsy (>1 seizure/month or >2 medication changes last 6 months)
7. Any TMS or MRI contraindication including implanted electronic devices
8. Botox, orthopedic surgery, or other invasive therapy in past 12 months
9. Constraint, brain stimulation or other modulatory therapy in past 6 months

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Assisting Hand Assessment (AHA) at 8 weeks | 8 weeks
  This is the established standard for the objective quantification of bilateral hand function in children with hemiparetic CP.This Rasch-built evaluation carries the strongest evidence of inter-rater, intra-rater, and test-retest reliabilities, test-validity, and responsiveness to change for bimanual tasks in children within our age range For more details about this measures please refer to the published literature.

SECONDARY OUTCOMES:
tDCS Safety and Tolerability evaluation (TST) | Each day following the tDCS treatment (10x)
  Adapted from a published safety consensus statements and child-friendly tolerability evaluations for non-invasive brain stimulation. Measure will capture all possible adverse events including severity and duration, rank tDCS sessions across common childhood experiences, and evaluate sham effectiveness. For more details about this measures please refer to the published literature.
Change from baseline in the Canadian Occupational Performance Measure (COPM) at 1 week | Baseline, 1 week
  Individualized, family-centered tool identifying child and family-perceived difficulties in self-care, productivity (school), and activities. OT-guided goal setting scores 3-5 individualized, realistic goals and ranks them on a scale of 1-10 for both satisfaction and performance. The same assessor applies the tool at post follow-ups without reminding the subject of previous scores. Such subjective measures are highly clinically relevant to assess perceived gains in children. COPM is validated for our population.
Change from baseline in the Canadian Occupational Performance Measure (COPM) at 8 weeks | 8 weeks
  Individualized, family-centered tool identifying child and family-perceived difficulties in self-care, productivity (school), and activities. OT-guided goal setting scores 3-5 individualized, realistic goals and ranks them on a scale of 1-10 for both satisfaction and performance. The same assessor applies the tool at post follow-ups without reminding the subject of previous scores. Such subjective measures are highly clinically relevant to assess perceived gains in children. COPM is validated for our population.

OTHER OUTCOMES:
Change from baseline function in the Jebsen Taylor Test of Hand Function (JTTHF) at 1 week | Baseline, 1 week
  Standardized timed test of unimanual upper extremity functional activities evaluating efficiency of movement. For more details about this measures please refer to the published literature.
Change in grip and pinch strength (GS, PS) (bilateral) at 1 week from baseline | Baseline, 1 week
  Simple measures of motor power, quantifiable with hand dynamometer and pinch meter. Main function is independent assessment of UNAFFECTED hand function to ensure no decline in function.
Change from baseline using the Box and blocks and Purdue pegboard tests daily during the trial | Baseline, daily during trial at start and end of session (20x)
  Box and blocks evaluates manual dexterity with a quick, functional relevant test with robust range applicable to this age range. Main purpose is to gauge daily motor learning effects. The Purdue pegboard test will serve a similar function with comparability to recent pediatric CIMT studies (not performed daily).
Change from baseline in the Melbourne Assessment of Unilateral Upper Limb Function (MAUULF) at 1 week | Baseline, 1 week
  Validated, criterion-referenced unimanual functional measure designed to detect therapeutic change in children with hemiparetic CP. High reliabilities and construct validity. For more details about this measures please refer to the published literature.
Change from baseline in the Quality of Life (QoL) assessment at 1 week | Baseline, 1 week
  Functional improvements may not correlate with health related QoL, necessitating evaluation in clinical trials. The CP QOL-Child is a psychometrically sound, condition specific instrument for children with CP (age 4-12). The Pediatric Quality of Life Inventory CP Module (PedsQL-CP) is condition specific and validated for child self-report (age 5-18) and will be completed by all participants. These tools will evaluate social and emotional well-being, participation, school activities, access to services, pain and feelings about disability, and family health.
Change from baseline in TMS Neurophysiology at 1 week | Baseline, 1 week
  Single and paired pulse TMS paradigms will evaluate subject motor neurophysiology including the following parameters from stroke and non-stroke hemispheres: RMT, AMT, stimulus-response curves, SICI, ICF, LICI, IHI, cSP, iSP.
Pre and post intervention Advanced Neuroimaging | Baseline, 1 week
  Standardized 3T MR protocol will be applied including anatomical volumetrics, task fMRI (affected, unaffected, and bimanual hand activations), resting state fMRI (primary outcome is M1 laterality index), diffusion tensor imaging (primary outcome is CST FA ratio) and bilateral M1 MR spectroscopy.
Change from baseline function in the Jebsen Taylor Test of Hand Function (JTTHF) at 8 weeks | 8 weeks
  Standardized timed test of unimanual upper extremity functional activities evaluating efficiency of movement. For more details about this measures please refer to the published literature.
Change in grip and pinch strength (GS, PS) (bilateral) at 8 weeks from baseline | 8 weeks
  Simple measures of motor power, quantifiable with hand dynamometer and pinch meter. Main function is independent assessment of UNAFFECTED hand function to ensure no decline in function.
Change from baseline using the Box and blocks and Purdue pegboard at 8 weeks | 8 weeks
  Box and blocks evaluates manual dexterity with a quick, functional relevant test with robust range applicable to this age range. Main purpose is to gauge daily motor learning effects. The Purdue pegboard test will serve a similar function with comparability to recent pediatric CIMT studies (not performed daily).
Change from baseline in the Melbourne Assessment of Unilateral Upper Limb Function (MAUULF) at 8 weeks | 8 weeks
  Validated, criterion-referenced unimanual functional measure designed to detect therapeutic change in children with hemiparetic CP. High reliabilities and construct validity. For more details about this measures please refer to the published literature.
Change from baseline in the Quality of Life (QoL) assessment at 8 weeks | 8 weeks
  Functional improvements may not correlate with health related QoL, necessitating evaluation in clinical trials. The CP QOL-Child is a psychometrically sound, condition specific instrument for children with CP (age 4-12). The Pediatric Quality of Life Inventory CP Module (PedsQL-CP) is condition specific and validated for child self-report (age 5-18) and will be completed by all participants. These tools will evaluate social and emotional well-being, participation, school activities, access to services, pain and feelings about disability, and family health.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kirton, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Kirton A, Ciechanski P, Zewdie E, Andersen J, Nettel-Aguirre A, Carlson H, Carsolio L, Herrero M, Quigley J, Mineyko A, Hodge J, Hill M. Transcranial direct current stimulation for children with perinatal stroke and hemiparesis. Neurology. 2017 Jan 17;88(3):259-267. doi: 10.1212/WNL.0000000000003518. Epub 2016 Dec 7. PMID 27927938
- See also: Program website — http://www.perinatalstroke.ca